CLINICAL TRIAL: NCT02724228
Title: A Phase 2, Open-Label, Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of BMN 111 in Children With Achondroplasia
Brief Title: A Study to Evaluate Long-Term Safety, Tolerability, & Efficacy of BMN 111 in Children With Achondroplasia (ACH)
Acronym: ACH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-205; 2015-004004-30 (EudraCT Number)
Record Dates: First submitted 2016-02-12; First posted 2016-03-31 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; Dwarfism; Bone Diseases, Developmental; Bone Diseases
MeSH Terms: conditions — Achondroplasia; Dwarfism; Bone Diseases, Developmental; Bone Diseases | interventions — vosoritide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMN 111 - Subcutaneous Injection (Experimental): 111-205 is an open-label, extension study. Subjects receive the same stable dose of BMN 111 received upon completion of the 111-202 study, initially up to 30 μg/kg. BMN 111 will be administered by weight-band dosing regimen.
  Interventions: Drug: BMN 111

INTERVENTIONS:
Drug: BMN 111 — BMN 111 will be administered subcutaneously daily.
  Other Names: Modified recombinant human C-type natriuretic peptide; Vosoritide

SUMMARY:
This is a Phase 2, Open-Label, Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of BMN 111 in Children with Achondroplasia. The primary objective is to evaluate the long-term safety and tolerability of daily SC injections of BMN 111 in children with ACH who have completed two years of treatment in the 111-202 study.

ELIGIBILITY:
Inclusion Criteria:

* Have completed 24 months of BMN 111 treatment in Study 111-202.
* Parent(s) or guardian(s) are willing and able to provide written, signed informed consent. Subjects under the age of majority are willing and able to provide written assent (if required). Subjects who reach the age of majority in their country will be asked to provide their own written consent upon reaching the legal age of majority.
* If sexually active, willing to use a highly effective method of contraception while participating in the study.
* Females >= 10 years old or who have started menses must have a negative pregnancy test at baseline and be willing to have additional pregnancy tests during the study
* Willing and able to perform all study procedures as physically possible
* Parents/caregivers willing to administer daily injections to the subjects and complete the required training.

Exclusion Criteria:

* Requires any investigational agent prior to completion of study period.
* Have a condition or circumstance that, in the view of the Investigator, places the subject at high risk for poor treatment compliance or for not completing the study.
* Concurrent disease or condition that, in the view of the Investigator, would interfere with study participation or safety evaluations for any reason.
* Permanently discontinued BMN 111 during the 111-202 study.
* Subject is pregnant at Baseline visit or planning to become pregnant (self or partner) at any time during the study.
* Current chronic therapy with restricted medications.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Until near final adult height is reached, and up to at least 16 years of age for females and 18 years of age for males, whichever occurs later
  * Number of study participants with treatment-emergent adverse events.
  * Number of study participants with treatment-emergent serious adverse events

SECONDARY OUTCOMES:
Growth Velocity [Efficacy] | Until near final adult height is reached
  Annualized growth velocity (cm/yr)
Growth Parameters (Efficacy) | Until near final adult height is reached, and up to at least 16 years of age for females and 18 years of age for males, whichever occurs later
  Height standard score (Z-score)
Body Proportions (Efficacy) | Until near final adult height is reached, and up to at least 16 years of age for females and 18 years of age for males, whichever occurs later
  Upper-to-lower body segment ratio
Final Adult Height | Up to at least 16 years of age for females and 18 years of age for males
  Height at the age of 16 years for females and 18 years for males

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (9):
- United States (6):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Ann and Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins McKusick - Institute of Genetic Medicine, Baltimore, Maryland
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Institut Necker, Paris, France
- Guys & St. Thomas NHS Foundation Trust Evelina Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi Y, Chan ML, Mould DR, Larimore K, Fisheleva E, Cherukuri A, Day J, Savarirayan R, Irving M, Bacino CA, Hoover-Fong J, Ozono K, Mohnike K, Wilcox WR, Bober MB, Henshaw J. Development of a Weight-Band Dosing Approach for Vosoritide in Children with Achondroplasia Using a Population Pharmacokinetic Model. Clin Pharmacokinet. 2024 May;63(5):707-719. doi: 10.1007/s40262-024-01371-6. Epub 2024 Apr 23. PMID 38649657
- [Derived] Savarirayan R, Irving M, Bacino CA, Bostwick B, Charrow J, Cormier-Daire V, Le Quan Sang KH, Dickson P, Harmatz P, Phillips J, Owen N, Cherukuri A, Jayaram K, Jeha GS, Larimore K, Chan ML, Huntsman Labed A, Day J, Hoover-Fong J. C-Type Natriuretic Peptide Analogue Therapy in Children with Achondroplasia. N Engl J Med. 2019 Jul 4;381(1):25-35. doi: 10.1056/NEJMoa1813446. Epub 2019 Jun 18. PMID 31269546